CLINICAL TRIAL: NCT06732232
Title: A Dose Escalating Study of CD19/CD22/BCMA Three Targets Autologous Chimeric Antigen Receptor T (CAR-T) Cell Therapy in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: A Dose Escalating Study of CD19/CD22/BCMA CAR-T Therapy in Relapsed/ Refractory Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZE2204-B-01
Record Dates: First submitted 2024-11-28; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Relapsed; Refractory; Multiple Myeloma
Keywords: relapsed/refractory multiple myeloma; CAR-T; CD19; CD22; BCMA
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/CD20/BCMA CAR-T cells therapy (Experimental): CD19/CD20/BCMA CAR T cells Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of CD19/CD20/BCMA CAR T cells. Cyclophosphamide and fludarabine will be given from day-5 to day-3 before the infusion for lymphodepletion. On day0 subjects will receive one dose treatment with CD19/CD20/BCMA CAR T cells by intravenous (IV) injection
  Interventions: Drug: CD19/CD20/BCMA CAR-T

INTERVENTIONS:
Drug: CD19/CD20/BCMA CAR-T — CD19/CD20/BCMA CAR T therapy

SUMMARY:
This is a single arm, open-label, dose escalation clinical study to evaluate the safety and tolerability of autologouschimeric antigen receptor T (CAR-T) cells targeting CD19/CD22/BCMA in patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a single arm, open-label, dose escalation investigator initiated (IIT) study, the primary objective is to evaluate the safety and tolerability of CD19/ CD22/BCMA CAR-T therapy in patients with relapsed/refractory multiple myeloma, and determine the maximum tolerated dose (MTD). For the secondary objectives,pharmacokinetics(PK), survival of CAR-T cells in vivo,pharmacodynamics (PD) and efficacy in R/R MM will be evaluated.

This study flow comprises of a screening phase( 30 to10 days prior to infusion), apheresis phase (9 to 8 days prior to infusion), lymphodepletion phase (5 to 3 days prior to infusion) , infusion of CD19/CD22/BCMA CAR-T cells on Day0, DLT assessments phase (from Day1 to Day 28) and post- treatment follow-up phase (Day 29 and up to end of the study).

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria in order to be enrolled:

  1. Understand and voluntarily sign an informed consent form (ICF) before conducting any research related evaluations/procedures;
  2. Age range: 18-75 years old;
  3. Expected survival period is not less than 12 weeks;
  4. ECOG score ≤ 2 points;
  5. The bone marrow flow cytometry results showed positive BCMA antigen (including weak positive, moderate positive, and strong positive);
  6. According to the IMWG criteria, a diagnosis of multiple myeloma with measurable lesions must meet at least one of the following criteria:

     1. Serum M protein (SPEP) ≥ 5g/L
     2. 24-hour urinary M-protein excretion rate ≥ 0.2g (200mg)
     3. Serum free light chain (sFLC) ≥ 100 mg/L and abnormal free light chain ratio
     4. The ratio of primitive plasma cells to immature plasma cells in bone marrow cytology examination is greater than 5%, or the flow cytometry detection of monoclonal plasma cells is greater than 5%
  7. Those who have received treatment with at least three different mechanisms of action (including anti-CD38 monoclonal antibodies, protease inhibitors, immunosuppressants, etc.) but have failed, and have experienced relapse (within 12 months), difficulty in treatment, or intolerance to the last line treatment regimen, including primary difficulty in treatment (subjects who have not achieved minimal remission [MR] or developed disease progression [PD] during treatment) or secondary difficulty in treatment (subjects who develop disease progression within 60 days after completion of treatment);
  8. There is no significant abnormality in lung function, and the oxygen saturation is greater than 92% in the absence of oxygen inhalation;
  9. The blood biochemistry test results meet the following criteria:

     1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
     2. Total bilirubin ≤ 1.5 × ULN
     3. 24-hour serum creatinine clearance rate ≥ 30 mL/min
     4. Lipase and amylase ≤ 2 × ULN
  10. The blood routine test meets the following criteria:

      1. Lymphocyte count>0.5 × 10 ^ 9/L
      2. Neutrophil count ≥ 1.0 × 10 ^ 9/L
      3. Hemoglobin ≥ 60g/L
      4. Platelets ≥ 40 × 10 ^ 9/L
  11. Men with fertility and women of childbearing age must agree to use effective contraceptive measures from the signing of the informed consent form until 2 years after the use of the study drug. Women of childbearing age include premenopausal women and women within 2 years after menopause. The blood pregnancy test for women of childbearing age must be negative during screening.

Exclusion Criteria:

* Any of the following situations cannot be selected as a subject:

  1. Asymptomatic (smoking type) multiple myeloma;
  2. Multiple myeloma with only extramedullary lesions present;
  3. Plasma cell leukemia;
  4. Merge amyloidosis;
  5. Central nervous system (CNS) metastasis, leptomeningeal disease, or metastatic central compression;
  6. Pregnancy or lactation period;
  7. Individuals who are HBsAg positive or HBcAb positive, unless HBV-DNA is less than 100 IU/ml or below the minimum detectable value; Individuals who are positive for hepatitis C virus (HCV) antibodies and HCV-RNA; Individuals who are HIV antibody positive; Individuals who are positive for syphilis specific antibodies and have a positive TRUST (toluidine red unheated serum test) test; Individuals who test positive for Cytomegalovirus (CMV) DNA;
  8. Cardiovascular diseases with clinical significance, including any of the following:

     1. QT interval (QTcF) after heart rate correction:>470 milliseconds;
     2. New York Heart Association Grade II and above heart failure;
     3. Left ventricular ejection fraction (LVEF) ≤ 50%;
     4. Poorly controlled hypertension (systolic blood pressure ≥ 150 mm Hg and/or diastolic blood pressure ≥ 95 mm Hg)
     5. Arrhythmias that have clinical significance or require antiarrhythmic treatment (such as persistent ventricular tachycardia, ventricular fibrillation, apical torsion tachycardia, and complete left bundle branch block);
  9. Has experienced unstable angina or acute myocardial infarction within the 6 months prior to signing the ICF;
  10. Previously received any anti-CD45 or anti-CD3 treatment;
  11. Individuals who are allergic to any of the components of the drugs used in this study, including but not limited to Qing Lin drugs (cyclophosphamide, fludarabine), etc;
  12. Received any investigational drug or systemic anti-tumor treatment within 4 weeks (or 5 half lives of the drug, whichever the researcher deems more appropriate) prior to single collection;
  13. History of other primary malignant tumors within 5 years prior to treatment, except for the following situations:

      1. Fully treat cured cervical carcinoma in situ;
      2. Localized basal cell carcinoma or squamous cell carcinoma of the skin;
  14. Any uncontrolled active infection within 4 weeks prior to single collection requires parenteral antibiotics, antiviral or antifungal treatment;
  15. Individuals with a history of active pulmonary tuberculosis infection within one year prior to single sampling (excluding subjects with a history of active pulmonary tuberculosis infection more than one year ago who, according to the researcher's judgment, currently have no evidence of active pulmonary tuberculosis);
  16. Accompanying or having a history of interstitial lung disease or interstitial pneumonia;
  17. Subjects who receive autologous hematopoietic stem cell transplantation (ASCT) within 8 weeks of signing the ICF, or who plan to undergo ASCT during the study period;
  18. Subjects who have received allogeneic stem cell therapy in the past; The researchers believe that complications or other conditions in the subjects may affect their compliance with the protocol or make them unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-12-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | [Time Frame: Day0-Day28]
  Safety
Maximum tolerated dose (MTD) | [Time Frame: Day0-Day28]
  Evaluate the incidence, severity, and correlation of SAE Tolerability

SECONDARY OUTCOMES:
Maximum Plasma Concentration(Cmax) | [Time Frame: Day0-Day28#Day0-undetectable for CAR positive T cells]
  Pharmacokinetics(PK)
Maximum Plasma Concentration Time (Tmax) | [Time Frame: Day0-Day28#Day0-undetectable for CAR positive T cells]
  Pharmacokinetics(PK)
Area Under Curve (AUC) | [Time Frame: Day0-Day28#Day0-undetectable for CAR positive T cells]
  Pharmacokinetics(PK)
CAR positive T cells | [Time Frame: Day0-Day28#Day0-undetectable for CAR positive T cells]
  Pharmacokinetics(PK)
Cytokines ( IL(interleukin)-2） | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
Cytokines ( IL(interleukin)-4） | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
Cytokines ( IL(interleukin)-6） | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
Cytokines ( IL(interleukin)-8） | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
Cytokines ( IL(interleukin)-10） | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
Cytokines ( IL(interleukin)-15） | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
IFN(interferon)-γ | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
TNF(tumor necrosis factor)-α | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
MCP( monocyte chemoattractant protein)-1) | [Time Frame:Day0-Day28]
  Pharmacodynamics (PD)
Overall survival (OS) | [Time Frame: Day28,Month2,Month3,Month6,Month9,Month12,Month15,Month18,Month21,Month24]
  Based on the analysis of MRD negative rate by researchers according to IMWG standards
Progression-free survival (PFS) | [Time Frame: Day28,Month2,Month3,Month6,Month9,Month12,Month15,Month18,Month21,Month24]
  Based on the analysis of MRD negative rate by researchers according to IMWG standards
Minor residual diseases(MRD) | [Time Frame: Day28,Month2,Month3,Month6,Month9,Month12,Month15,Month18,Month21,Month24]
  Based on the analysis of MRD negative rate by researchers according to IMWG standards

CONTACTS AND LOCATIONS:
Overall Officials: Jinxing Lou, Principal Investigator — China, Shanghai Mengchao Cancer Hospital
Locations (1):
- China, Shanghai Mengchao Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No